CLINICAL TRIAL: NCT05073822
Title: A Phase III, Randomised, Single-site Trial on the Minimisation of Immunosuppression In Elderly Renal Transplant Recipients.
Brief Title: NOMINATE/ Minimisation of Immunosuppression in Kidney Transplantation
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding not secured
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 140986
Record Dates: First submitted 2021-09-16; First posted 2021-10-12 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Renal Transplant Rejection; Renal Transplant Infection
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: The investigators propose to conduct the study in two phases. Phase I will randomise renal transplant recipients over the age of 60yrs to either standard of care Immunosuppression (SOC-IS) or minimised immunosuppression (Min-IS) therapy, with monitoring of plasma dd-cfDNA levels over the first post-transplant year.
  There will be different target drug levels for tacrolimus: SOC-IS target levels of 8-12ng/ml in the first 3 months, 6-8ng/ml in months 4-12 and 4-8ng/ml after the 1st year; Min-IS levels 6-8ng/ml for first 3 months and 4-8ng/ml in months 4-12, For mycophenolate there will be two doses used: SOC-IS dose starting at 2g/day for 1 month, then 1.5mg/day between months 2-12, and then 1g/day after the 1st year; for Min-IS 1.5g/day in the first month and then 1g/day until 1 year post-transplantation. Outcomes will be assessed by the end of year 1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard of care Immunosuppression (SOC-IS) therapy (Other): serum tacrolimus level : target tacrolimus levels 8-12ng/ml in the first 3 months target tacrolimus levels 6-8ng/ml in months 4-12 target tacrolimus level 4-8ng/ml after the 1st year
  Mycophenolate mofetil dose :
  2g/day for 1 month 1.5mg/day between months 2-12
  1g/day after the 1st year
  Interventions: Drug: Tacrolimus
- minimised immunosuppression (Min-IS) therapy (Other): serum tacrolimus level : target tacrolimus levels 6-8ng/ml for first 3 months target tacrolimus levels 4-8ng/ml in months 4-12.
  Mycophenolate mofetil dose:
  1.5g/day in the first month
  1g/day until 1 year post-transplantation
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — reduction of both standard Tacrolimus & Mycophenolate mofetil does in one arm
  Other Names: Tacrolimus, Mycophenolate mofetil

SUMMARY:
Kidney transplantation provides the optimal form of kidney replacement therapy for the majority of people with end-stage kidney disease, and has now become the commonest form of kidney replacement therapy. However, donor and recipient demographics have changed considerably over the past few decades: increasingly older donor kidneys are transplanted into progressively older recipients with greater comorbidities. Increasing age remains a major risk factor for death after kidney transplantation, with the commonest causes of deaths for recipients aged 70 and over being cardiovascular, infection, and malignancies. Immunosuppressant drugs which are critical for the maintenance of the transplanted organ can contribute to increased morbidity and mortality, by direct effects or through lowered immunity predisposing to infection. Cytomegalovirus (CMV) is one of the most common opportunistic infections that affects renal transplant patient outcome and can be monitored prospectively. Hence, minimising immunosuppression, especially in older recipients, may result in better graft and patient outcomes as many side-effects are dose dependant. However, to date drug doses have never been adjusted based on age, despite significant changes that occur to immune responsiveness as patients grow older. In addition , researchers have not had a biomarker to help define appropriate immunosuppressive levels for each individual.

The investigators therefore aim to study the effect of reducing the target immunosuppression drug levels( of tacrolimus and mycophenolate) in kidney transplant recipients >60 years, using CMV viraemia as a main outcome measure, and investigating rates of rejection and development of de novo donor-specific anti-HLA antibodies. The investigators will assess the clinical utility of donor-derived cell free DNA (dd-cfDNA) as a means to guide immunosuppression minimisation. The investigators propose that the use of lower doses of immunosuppression will result in fewer infection-related complications, translating to improved patient outcomes. The research will be carried out in kidney transplant centres where prospective CMV monitoring is practiced.

DETAILED DESCRIPTION:
Older kidney transplant recipients are at increased risk of infection and death from infectious causes compared to younger transplant recipients, and despite knowledge of age related immunological changes, the immunosuppressive protocol for older recipients was not yet adjusted. Our provisional data suggest that standard dose immunosuppression in the older patients results in more infections and fewer rejection episodes. Achieving a better balance by reducing risk of infection would be highly desirable. Defining age-specific target drug levels and doses should therefore be tested in a formal trial to establish its validity.

Transplant recipients are especially at risk from viral and opportunistic infections; CMV is a particular problem, as infections can be both donor-derived or due to re-activation of latent virus in the recipient. In the transplant population, CMV infection can cause significant morbidity, including bone marrow suppression, pneumonitis, colitis, retinitis and encephalitis, and as a consequence, increased mortality. However, as this will be measured prospectively, it can also be utilised as a marker of the degree of ( over) immunosuppression in our patients.

There are no current recommendations regarding optimal dose or target drug levels, and importantly, no age-specific standards. This trial could provide some specific recommendations.

There is an increasing body of evidence that demonstrates age-related changes to the immune system, termed immunosenescence, characterized by reduced responsiveness to both newly and previously encountered antigens. In transplantation, it is thought that such immunosenescence may influence both the immune response of the recipient and the immunogenicity of the donor organ. Understanding if this is in any way related to physical frailty may be helpful in informing patients of risk of transplantation.

Donor-derived cell-free DNA (dd-cfDNA) detected in the plasma of transplant recipients has been increasingly reported as a noninvasive biomarker of acute rejection(AR)-with transplant organ damage leading to release of more of the donor DNA into the bloodstream. A recent systematic review showed that all but one of 48 relevant studies reported significant elevations of dd-cfDNA at the time of biopsy-proven AR (BPAR), with successful treatment of AR resulting in restoration of dd-cfDNA levels back to baseline. Furthermore, a rise in dd-cfDNA can be detected before the clinical manifestations of rejection, with elevated levels seen up to a month or more before diagnosis of BPAR in some studies. Using the stability of the marker( a lack of rise) as a means of customising therapy has not been attempted, and our study could provide the rationale for this strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be first time adult recipients of either a deceased or living donor kidney transplant.
2. Participant must be a recipient of a single organ transplant only.
3. Participant must be above the age of 60 years.
4. Participant must have a negative screen for donor-specific antibody prior to transplantation (MFI<2000).

Exclusion Criteria:

1. Recipients of a transplant who are highly sensitised (cRF >85%).
2. Inability to participate in frequent monitoring of renal transplant function and clinical visits (every 4 weeks) during dd-cfDNA monitoring and IS minimisation.
3. Participants with immune-mediated renal disease in which IS minimisation is inadvisable.
4. EBV negative recipient (as IS minimisation is part of standard protocol)
5. Inability to comply with study directed treatment

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2027-02-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
CMV viraemia | one year
  Incidence of CMV viraemia as defined as any detectable virus by (PCR) above the threshold of 200 copies/ml in 1st year

SECONDARY OUTCOMES:
Incidence of biopsy-proven acute rejection | 1 year
  1.Incidence of biopsy-proven acute rejection by 12 months after randomization

IPD SHARING:
Plan to Share IPD: No